CLINICAL TRIAL: NCT05943886
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled, Single and Multiple Dose Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HEC88473 Injection in Healthy Subjects, Obese Subjects and T2DM Subjects
Brief Title: A Phase 1 Study of HEC88473 Injection in Healthy Subjects, Obese Subjects and T2DM Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongguan HEC Biopharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC88473-DM-101
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Healthy Subjects; Obesity; T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Single dose of 0.5 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 0.5 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 1.7 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 1.7 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 5.1 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 5.1 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Obese subjects, receiving a single dose of 5.1 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 10.2 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 10.2 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 17.0 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 17.0 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 25.5 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 25.5 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 35.7 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 35.7 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 47.6 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 47.6 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 62.9 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 62.9 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 81.6 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 81.6 mg HEC88473 (N=8) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 5.1 mg HEC88473 (Experimental): T2DM subjects, receiving a weekly dose of 5.1 mg HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 15.3 mg HEC88473 (Experimental): T2DM subjects, receiving a weekly dose of 15.3 mg HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 30.6 mg HEC88473 (Experimental): T2DM subjects, receiving a weekly dose of HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  The 30.6 mg cohort was administered by titration.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 45.9 mg HEC88473 (Experimental): T2DM subjects, receiving a weekly dose of HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  The 45.9 mg cohort was administered by titration.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 68.0 mg HEC88473 (Experimental): T2DM subjects, receiving a weekly dose of HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  The 68.0 mg cohort was administered by titration.
  Interventions: Drug: HEC88473 injection; Drug: Placebo

INTERVENTIONS:
Drug: HEC88473 injection — HEC88473 will be provided as a 17 mg/mL solution and will be administered by subcutaneous injection in the abdomen.
Drug: Placebo — Placebo will be administered by subcutaneous injection in the abdomen.

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, escalating single-dose and multiple-dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HEC88473 injection in healthy subjects, obese subjects and subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This study is divided into two parts, Part A is an escalating single-dose study in healthy subjects and obese subjects, and Part B is an escalating multiple-dose study in subjects with T2DM.

ELIGIBILITY:
Inclusion Criteria:

Part A

1. Males or females, between 18 and 45 years of age, inclusive, at screening.
2. Body weight ≥ 50 kg for males and body weight ≥ 45 kg for females. 18≤body mass index (BMI)<28 kg/m2 for nonobese subjects and 28≤BMI≤45 kg/m2 for obese subjects.

Part B

1. Males or females, between 18 and 65 years of age, inclusive, at screening.
2. 24 kg/m2≤BMI≤35 kg/m2.
3. Subjects diagnosed with T2DM, newly diagnosed subjects at screening, or treated with diet and exercise alone within 3 months before screening and still have poor blood glucose control, or treated with a stable dose of metformin for ≥ 3 months before screening.
4. 7.0%≤ HbA1c ≤10.5% at screening.

Exclusion Criteria:

Part A

1. Smoked more than 5 cigarettes per day within 3 months before the study.
2. Immunization with a live attenuated vaccine or coronavirus vaccination within 1 month prior to screening or planned vaccination during the course of the study.
3. Positive alcohol breath test result or positive urine drug screen.
4. Blood donation (> 300 mL) or massive blood loss (> 400 mL) within 3 months before screening.

Part B

1. Have type 1 diabetes mellitus.
2. Have had ≥1 episode of severe hypoglycemia within 6 months before screening, or history of recurrent hypoglycemia (history of hypoglycemia more than 3 times in 3 months).
3. Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine aminotransferase (ALT) level >5 times the upper limit of the reference range at screening.
4. Have serum calcitonin ≥20 ng/L at screening.
5. Have a personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2; or have hereditary diseases that can easily induce MTC.
6. Fasted triglycerides > 5.7 mmol/L at screening. If the patient is on lipid-lowering therapies, doses must be stable for 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) after a single dose of HEC88473 | Baseline to day 15
  Adverse Events (AEs)
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) after multiple dose of HEC88473 | Baseline to day 43
  Adverse Events (AEs)
Cmax | Predose and postdose 4、8、10、12、14、24、48、72、96、168、216、336 hours
  Maximum observed serum concentration of HEC88473
AUC | Predose and postdose 4、8、10、12、14、24、48、72、96、168、216、336 hours
  Area under the serum concentration-time curve (AUC)

SECONDARY OUTCOMES:
OGTT | Day-1, Day3 and Day 7
  Oral glucose tolerance test
Change from baseline of Adiponectin at day 38 | Baseline to day 38
  Adiponectin
Fasting lipid concentration | Baseline to day 43
  Fasting lipid concentration
Change from baseline of HbA1c at day 38 | Baseline to day 38
  HbA1c
Assessment of the incidence of anti drug antibodies (ADA) developed against HEC88473 after dosing | Baseline to day 43
  anti drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Zhang H, Li Q, Chen H, Guo L, Li J, Xie C, Yan J, Ding Y. First-in-Human Study on Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Escalating Doses of HEC88473, a Novel Dual GLP-1 and FGF21 Receptor Agonist in Healthy and Obese Chinese Subjects. BioDrugs. 2025 May;39(3):477-486. doi: 10.1007/s40259-025-00715-3. Epub 2025 Apr 3. PMID 40175670
- [Derived] Xiang L, Wang G, Zhuang Y, Luo L, Yan J, Zhang H, Li X, Xie C, He Q, Peng Y, Chen H, Li Q, Li X, Guo L, Lv G, Ding Y. Safety and efficacy of GLP-1/FGF21 dual agonist HEC88473 in MASLD and T2DM: A randomized, double-blind, placebo-controlled study. J Hepatol. 2025 Jun;82(6):967-978. doi: 10.1016/j.jhep.2024.12.006. Epub 2024 Dec 19. PMID 39709140